CLINICAL TRIAL: NCT05611203
Title: Molecular Detection of SARS-CoV-2 From Oropharyngeal Swabs Performed With or Without Specimen Collection From the Palatine Tonsils - a Multicenter Randomized Controlled Trial
Brief Title: Should Palatine Tonsils be Included in the Oropharyngeal Swab for SARS-CoV-2 Molecular Testing?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Tobias Todsen, Consultant, Associate Prof, Rigshospitalet, Denmark
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-22022937
Record Dates: First submitted 2022-11-03; First posted 2022-11-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: SARS-CoV Infection; Coronavirus; Corona Virus Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oropharyngeal swab only including the posterior oropharyngeal wall (Experimental): An Oropharyngeal swab is performed with the collection of specimens from the posterior oropharyngeal wall only
  Interventions: Procedure: An Oropharyngeal swab
- Oropharyngeal swab including the posterior oropharyngeal wall and both palatine tonsils (Experimental): An Oropharyngeal swab is performed with the collection of specimens from the posterior oropharyngeal wall and both palatine tonsils
  Interventions: Procedure: An Oropharyngeal swab

INTERVENTIONS:
Procedure: An Oropharyngeal swab — An Oropharyngeal swab performed for diagnostic purposes

SUMMARY:
Citizens who undergo testing for COVID-19 at one of two Testcenters in Copenhagen Captial Region will be invited to participate in the study. The participants will be randomized to either an oropharyngeal swap including the palatine tonsils OR an oropharyngeal swap without the palatine tonsils for SARS-CoV-2 testing. The swabs will be sent to the clinical microbiology laboratory for SARS-CoV-2 detection using RT-PCR. The diagnostic accuracy and SARS-CoV-2 viral load will be compared. The participants will be asked to complete a questionnaire regarding their symptoms.

DETAILED DESCRIPTION:
We will include citizens referred for outpatient testing for COVID-19 who will be offered to participante in the study on a volunteer basis. Participants are all volunteers, who are attending the test facilities to obtain a PCR test. Participants are required to provide oral and written informed consent to participate before entering the study. The inclusion criterion is 18 years or more of age. Exclusion criteria are neck breathers (tracheostomy/laryngectomy patients).

The participants will be randomized to either an oropharyngeal swap including the palatine tonsils OR an oropharyngeal swap without the palatine tonsils for SARS-CoV-2 testing.

The swabs will be sent to the clinical microbiology laboratory for SARS-CoV-2 detection using RT-PCR as usual. The diagnostic accuracy and SARS-CoV-2 viral load will be compared using independent t-test. The participants will be asked to complete a questionnaire regarding their symptoms and the number of sick days. All data will be documented on-site in a secure web database (REDCap).

The primary outcome will be reported as:

• SARS-CoV-2 RNA by RT-PCR test result (positive, negative, inconclusive)

The secondary outcome will be reported as:

* SARS-CoV-2 RT-PCR cycle threshold (Ct) value
* Test discomfort on a 11-point NRS-scale
* Development of COVID-19 disease after testing
* SARS-CoV-2 detection rate for each healthcare worker
* Mallampati Score of participants being tested

ELIGIBILITY:
Inclusion Criteria:

* citizens referred for outpatient testing for COVID-19 in Valby and Hillerød COVID-19 TestCenter.

Exclusion Criteria:

* Age under 18 years
* neck breathers (tracheostomy/laryngectomy patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
RT-PCR results | Day 1
  The detection rate of SARS-CoV-2 RNA

SECONDARY OUTCOMES:
Sycle threshold (Ct) | Day 1
  SARS-CoV-2 RT-PCR cycle threshold (Ct) values
Inconclusive tests | Day 1
  Number of inconclusive RT-PCR tests results
Test discomfort | Day 1
  Self reported on a 11-point NRS-scale from 0 - 10 (with 10 being the worst imaginable discomfort)
Development of COVID-19 disease after testing | 1 month
  Online questionare about symptoms send by email
Test accuracy between healthcare workers | Day 1
  SARS-CoV-2 detection rate for each healthcare worker
Participants oropharynx anatomy | Day 1
  Mallampati Score of participants

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Hillerød Covid-19 Testcenter, Copenhagen, Hillerød
  - Valby, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided
Not decided

REFERENCES:
- [Derived] Hartvigsen B, Jakobsen KK, Benfield T, Gredal NT, Ersboll AK, Gronlund MW, Bundgaard H, Andersen MP, Steenhard N, von Buchwald C, Todsen T. Molecular Detection of SARS-CoV-2 From Throat Swabs Performed With or Without Specimen Collection From the Tonsils: Protocol for a Multicenter Randomized Controlled Trial. JMIR Res Protoc. 2024 Jun 12;13:e47446. doi: 10.2196/47446. PMID 38865190

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT05611203/Prot_SAP_ICF_000.pdf